CLINICAL TRIAL: NCT02412501
Title: A Clinical Evaluation of the Medtronic Resolute Onyx Zotarolimus-Eluting 2.0 mm Stent Resolute Onyx 2.0 mm Clinical Study
Brief Title: Medtronic Resolute Onyx 2.0 mm Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 5.0 - 26Mar2015
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device (Other): Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent System 2.0 mm Stent
  Interventions: Device: Resolute Onyx Stent - 2.0 mm

INTERVENTIONS:
Device: Resolute Onyx Stent - 2.0 mm — Clinical Evaluation of the Medtronic Resolute Onyx Zotarolimus-Eluting 2.0 mm Stent

SUMMARY:
The purpose of this trial is to assess the safety and efficacy of the Resolute Onyx Zotarolimus-Eluting Coronary Stent System for the treatment of de novo lesions in native coronary arteries that allows the use of a 2.0 mm diameter stent.

ELIGIBILITY:
Inclusion Criteria:

* Must be an acceptable candidate for percutaneous coronary intervention, stenting, & emergent coronary artery bypass graft (CABG) surgery
* Must have evidence of ischemic heart disease
* Must require treatment of either a) a single target lesion amenable to treatment with a 2.0 mm stent OR b) two target lesions located in separate target vessels, with at least one of the target lesions amenable to treatment with a 2.0 mm study stent
* Target lesion(s) must be de novo lesion(s) in native coronary artery(ies)

Exclusion Criteria:

* Known hypersensitivity or contraindication to aspirin, heparin and bivalirudin, thienopyridines, cobalt, nickel, platinum, iridium, chromium, molybdenum, polymer coatings (e.g. BioLinx) or a sensitivity to contrast media, which cannot be adequately pre-medicated
* History of an allergic reaction or significant sensitivity to drugs such as zotarolimus, rapamycin, tacrolimus, everolimus, or any other analogue or derivative
* History of a stroke or transient ischemic attack (TIA) within the prior 6 months
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Concurrent medical condition with a life expectancy of less than 12 months
* Currently participating in an investigational drug or another device trial that has not completed the primary endpoint
* Documented left ventricular ejection fraction (LVEF) < 30% at the most recent evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-04-06 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Price, MD, FACC, FSCAI, Principal Investigator — Scripps Green Hospital; Shigeru Saito, MD, Principal Investigator — Shonan Kamakura General Hospital
Locations (17):
- United States (17):
  - Scripps Green Hospital, La Jolla, California
  - Morton Plant Hospital, Clearwater, Florida
  - Saint John's Hospital, Springfield, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Barnes Jewish University, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - The Mount Sinai Medical Center, New York, New York
  - Saint Francis Hospital, Roslyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Medical Center, Fargo, North Dakota
  - University Hospitals Elyria Medical Center, Elyria, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - AnMed Health Medical Center, Anderson, South Carolina
  - Centennial Medical Center, Nashville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - East Texas Medical Center, Tyler, Texas

REFERENCES:
- [Derived] Price MJ, Saito S, Shlofmitz RA, Spriggs DJ, Attubato M, McLaurin B, Popma Almonacid A, Brar S, Liu M, Moe E, Mehran R. First Report of the Resolute Onyx 2.0-mm Zotarolimus-Eluting Stent for the Treatment of Coronary Lesions With Very Small Reference Vessel Diameter. JACC Cardiovasc Interv. 2017 Jul 24;10(14):1381-1388. doi: 10.1016/j.jcin.2017.05.004. PMID 28728650

RESULTS

PARTICIPANT FLOW:
Groups:
- Device: Medtronic Resolute Onyx Zotarolimus-Eluting Stent System >
  > Resolute Onyx Stent - 2.0 mm
Period: Overall Study
Arm/Group | Device
Started | 101
Completed | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Device: Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent System >
  > Clinical Evaluation of the Medtronic Resolute Onyx Zotarolimus-Eluting 2.0 mm Stent
Arm/Group | Device
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 82
  Black or African American | 3
  Asian | 15
  American Indian or Alaska Native | 1
Region of Enrollment [Number; unit: participants]
  United States | 86
  Japan | 15
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.0 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Target Lesion Failure at 12 Months Post-Procedure
Description: Target Lesion Failure at 12 months post-procedure, defined as Cardiac Death, Target Vessel Myocardial Infarction (Q wave or non-Q wave) or Target Lesion Revascularization by percutaneous or surgical methods.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Groups:
- Device: Medtronic Resolute Onyx Zotarolimus-Eluting Coronary Stent System 2.0 mm Stent >
  > Resolute Onyx Stent - 2.0 mm: Clinical Evaluation of the Medtronic Resolute Onyx Zotarolimus-Eluting 2.0 mm Stent
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 5

2. Secondary Outcome: Number of Participants With Cardiac Death at 12 Months Post Procedure
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 0

3. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TVMI) at 12 Months Post Procedure
Description: TVMI defined as Q Wave or non-Q Wave MI
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 3

4. Secondary Outcome: Number of Participants With a Major Adverse Cardiac Event at 12 Months Post Procedure
Time Frame: 12Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 5

5. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) at 24 Months Post Procedure
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 13

6. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) at 12 Months Post Procedure
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 5

7. Secondary Outcome: Number of Participants With Stent Thrombosis (ST) at 12 Months Post Procedure
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 0

8. Secondary Outcome: Number of Participants With Cardiac Death at 24 Months Post Procedure
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 2

9. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TVMI) at 24 Months Post Procedure
Description: TVMI defined as Q Wave or non-Q Wave MI
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 4

10. Secondary Outcome: Number of Participants With a Major Adverse Cardiac Event at 24 Months Post Procedure
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 14

11. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) at 24 Months Post Procedure
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 14

12. Secondary Outcome: Number of Participants With Stent Thrombosis (ST) at 24 Months Post Procedure
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 0

13. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF) at 36 Months Post Procedure
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 14

14. Secondary Outcome: Number of Participants With Cardiac Death at 36 Months Post Procedure
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 2

15. Secondary Outcome: Number of Participants With Target Vessel Myocardial Infarction (TVMI) at 36 Months Post Procedure
Description: TVMI defined as Q Wave or non-Q Wave MI
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 4

16. Secondary Outcome: Number of Participants With a Major Adverse Cardiac Event at 36 Months Post Procedure
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 15

17. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) at 36 Months Post Procedure
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 15

18. Secondary Outcome: Number of Participants With Stent Thrombosis (ST) at 36 Months Post Procedure
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 101
Participants | 0

ADVERSE EVENTS:
Time Frame: 36 months
Groups:
- 1. Onyx 2.0mm: Medtronic Onyx 2.0mm
Arm/Group | 1. Onyx 2.0mm
All-Cause Mortality (participants affected / at risk) | 3/101
Serious Adverse Events (participants affected / at risk) | 63/101
Other Adverse Events (participants affected / at risk) | 43/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Onyx 2.0mm (N=101)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)
Acute Left Ventricular Failure (Cardiac disorders) | 3 (3)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2)
Angina Pectoris (Cardiac disorders) | 3 (3)
Angina Unstable (Cardiac disorders) | 2 (2)
Anginal Equivalent (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (3)
Atrial Flutter (Cardiac disorders) | 2 (2)
Atrial Tachycardia (Cardiac disorders) | 1 (1)
Cardiac Aneurysm (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 11 (12)
Coronary Artery Stenosis (Cardiac disorders) | 5 (7)
Myocardial Ischaemia (Cardiac disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (2)
Eye Swelling (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastric Perforation (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 2 (2)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 2 (2)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Chest Pain (General disorders) | 5 (6)
Chills (General disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vascular Stent Stenosis (General disorders) | 6 (7)
Biliary Colic (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1)
Bronchitis Bacterial (Infections and infestations) | 2 (3)
Clostridium Difficile Colitis (Infections and infestations) | 2 (2)
Colon Gangrene (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Extradural Abscess (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (8)
Pneumonia Mycoplasmal (Infections and infestations) | 1 (1)
Post Procedural Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sepsis Syndrome (Infections and infestations) | 1 (1)
Staphylococcal Sepsis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (6)
Cartilage Injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 (1)
Plaque Shift (Injury, poisoning and procedural complications) | 2 (2)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (2)
Transplant Failure (Injury, poisoning and procedural complications) | 1 (1)
Traumatic Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Traumatic Renal Injury (Injury, poisoning and procedural complications) | 1 (1)
Haematocrit Decreased (Investigations) | 1 (1)
Haemoglobin Decreased (Investigations) | 1 (1)
Troponin Increased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oral Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oropharyngeal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous Cell Carcinoma Of The Oral Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 3 (3)
Cerebrovascular Accident (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Transient Ischaemic Attack (Nervous system disorders) | 2 (2)
Device Occlusion (Product Issues) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Bladder Outlet Obstruction (Renal and urinary disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Nephropathy Toxic (Renal and urinary disorders) | 1 (1)
Renal Cortical Necrosis (Renal and urinary disorders) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 1 (1)
Hypertensive Emergency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Intermittent Claudication (Vascular disorders) | 2 (2)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 2 (2)
Peripheral Artery Aneurysm (Vascular disorders) | 1 (1)
Peripheral Vascular Disorder (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Onyx 2.0mm (N=101)
Chest Pain (General disorders) | 15 (18)
Non-Cardiac Chest Pain (General disorders) | 6 (7)
Myocardial Necrosis Marker Increased (Investigations) | 7 (7)
Troponin I Increased (Investigations) | 6 (6)
Troponin Increased (Investigations) | 9 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (17)
Hypertension (Vascular disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2015-03-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT02412501/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT02412501/SAP_001.pdf